CLINICAL TRIAL: NCT00435448
Title: A Randomized Phase 3, Double-Blind, Placebo-Controlled Study of the Efficacy and Safety of Lonidamine for the Treatment of Symptomatic Benign Prostatic Hyperplasia
Brief Title: Study of the Efficacy and Safety of Lonidamine for the Treatment of Symptomatic Benign Prostatic Hyperplasia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Threshold Pharmaceuticals (Industry)
Collaborators: PRA Health Sciences (Industry)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: TH-CR-202
Record Dates: First submitted 2007-02-08; First posted 2007-02-15 (Estimated); Last update posted 2009-04-29 (Estimated); Status verified 2009-04

CONDITIONS: Benign Prostatic Hyperplasia; Enlarged Prostate
Keywords: Benign Prostatic Hyperplasia; BPH; Enlarged Prostate
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — lonidamine

INTERVENTIONS:
Drug: Lonidamine

SUMMARY:
The purpose of this study is to evaluate the efficacy of lonidamine (50mg, 150mg) compared to placebo in subjects with symptomatic BPH.

ELIGIBILITY:
Inclusion Criteria:

* Capable of understanding the purpose and risks of the study and sign a statement of informed consent
* Male 50-80 years of age
* Presence of LUTS (lower urinary tract symptoms) for at least 3 months
* Prostate volume measured by TRUS (transrectal ultrasound) > 30 cc
* Qmax < 15 mL/sec when measured by uroflowmetry (minimum of 125 mL must be voided)
* I-PSS (International prostate symptom score) > 12
* PSA > 1.0 ng/mL
* Must ensure and consent to use medically acceptable methods of contraception throughout the entire study with sexual partners of childbearing potential
* Able to comply with the prescribed treatment protocol and evaluations

Exclusion Criteria:

* Prior treatment for BPH with alpha-blockers and/or herbal supplements in the past 2 weeks (alpha-blockers and herbal supplements for the treatment of BPH are not allowed during the study). Prior treatment with 5-alpha-reductase inhibitors is allowed if discontinued at least 3 months prior to enrollment.
* Prior surgery of the prostate (except biopsies; subject is eligible to enroll one month after full recovery from prostate biopsy.)
* Current or past evidence of malignant disease of the prostate or prostatic intraepithelial neoplasia (for subjects with PSA between 4 - 10 ng/mL, prostate cancer must be ruled out to the satisfaction of the Principal Investigator. Subjects with PSA >10 ng/mL are excluded.)
* Active urinary tract infections (UTI)
* Active cardiac, renal or hepatic disease as evidenced by:

  1. Serum creatinine > 1.8 mg/dL
  2. ALT or AST > 2.5x the upper limit of normal at screen
  3. History of active myocardial infarction,unstable cardiac arrhythmias or stroke within 6 months prior to screening
  4. Uncontrolled congestive heart failure
* Uncontrolled diabetes mellitus (fasting blood glucose > 200 mg/dL)
* Use of systemic teriods for any reason (systemic steroid usage is not allowed during the study). Inhaled and/or topical steroids are allowed.
* Concurrent participation or participation in an investigational drug study within the past 30 days prior to screening
* Concomitant disease or condition that could interfere with the conduct of the study, or would in the opinion of the investigator,pose an unnaceptabele risk to the subject

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480
Dates: Start 2005-06; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
International prostate symptom score (I-PSS)

SECONDARY OUTCOMES:
Qmax on uroflowmetry
Post micturitional residue
Volume of the prostate
PSA

CONTACTS AND LOCATIONS:
Overall Officials: Peter Alken, MD, Principal Investigator — Fakultät für Klinische Medizin Mannheim
Locations (58):
- Germany (19):
  - Vivantes Klinikum am Urban, Klinik für Urologie, Berlin
  - ClinPharm International GmbH & Co KG--Chemnitz, Chemnitz
  - Universitätsklinik Köln, Klinik und Poliklinik für Urologie, Cologne
  - ClinPharm International GmbH & Co KG--Dresden, Dresden
  - niversitätsklinikum Carl Gustav Carus, Klinik und Poliklinik für Urologie, Dresden
  - Gemeinschaftspraxis Jacobi - Hellmis, Duisburg
  - ClinPharm International GmbH & Co KG--Frankfurt/Main, Frankfurt
  - ClinPharm International GmbH & Co KG--Gorlitz, Görlitz
  - Universitätsklinikum Hamburg-Eppendorf, Klinik und Poliklinik für Urologie, Hamburg
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Klinik für Urologie und Kinderurologie, Kiel
  - ClinPharm International GmbH & Co KG--Leipzig, Leipzig
  - ClinPharm International GmbH & Co KG--Magdeburg, Magdeburg
  - Urologische Universitätsklinik, Klinikum Mannheim gGmbH, Fakultät für Klinische Medizin Mannheim, Mannheim
  - Klinik für Urologie und Kinderurologie, Klinikum Marburg, Marburg
  - Klinikum der Universität München, Urologische Klinik und Poliklinik, München
  - Urologische Klinik und Poliklinik der Technischen Universität München, Klinikum Rechts der Isar, München
  - Urologische Klinik, Klinikum Landkreis Neumarkt i.d.Obf., Neumarkt
  - Klinik für Urologie, Eberhard-Karls-Universität Tübingen, Tübingen
  - Wuppertaler Gemeinschaftspraxis für Dermatologie, Gynäkologie und Urologie, Wuppertal
- Hungary (11):
  - Károlyi Sándor Hospital, Budapest
  - Semmelweis University, Budapest
  - Fővárosi Önkormányzat Jahn Ferenc Dél-Pesti Kórház, Budapest
  - Clinic of Urology, Debrecen
  - Dombóvári Szt. Lukács Egészségügyi Közhasznú, Dombóvár
  - Petz Aladár County Hospital, Győr
  - Kaposi Mór County Hospital, Kaposvár
  - Nagykanizsa Megyei Jogú Város Hospital, Nagykanizsa
  - Gróf Esterházy Kórház, Pápa
  - Dr. Bugyi István Hospital, Szentes
  - Saint Bobála Hospital, Tatabánya
- Italy (13):
  - A.O. Policlinico di Bari, Clinica Urologica I, Bari
  - A.O. Policlinico di Bari, Clinica Urologica, Bari
  - Ospedale S.Annunziata, Unità Operativa di Urologia, Florence
  - Università di Genova Ospedale S. Martino, Reparto Urologia, Genova
  - Ospedale S.Paolo, Cattedra di Urologia, Milan
  - Università Federico II, Clinica Urologica Edificio 5, Napoli
  - Azienda Ospedaliera S.Luigi di Orbassano, Reparto di urologia universitaria, Orbassano
  - Azienda Ospedaliera, Dipartimento di Urologia, Padua
  - A.O. Pliclinico Paolo Giaccone, U.O. Urologia con Litotrissia Extracorporea, Palermo
  - Azienda Ospedaliera Pisana, Dipartimento di Urologia 1, Pisa
  - Policlinico Sassarese, Istituto di Clinica Urologica, Sassari
  - Ospedale Maggiore S.Giovanni Battista, Istituto di Urologia, Torino
  - Ospedale S.Giovanni Bosco, Dipartimento di Urologia, Torino
- Poland (15):
  - Szpital Bielański, Oddział Urologii, Warsaw, Warszawa
  - Klinika Urologii AM w Białymstoku, Bialystok
  - Wojewódzki Szpital Specjalistyczny nr 4, Bytom
  - Gabinet Urologiczny, Gdansk
  - Specjalistyczna Praktyka Lekarska, Katowice
  - Szpital Specjalistyczny Oddzial Urologii, Kościerzyna
  - "Specjalista" Spółka z o. o., Kutno
  - Wojewódzki Szpital,Oddział i Poradnia Urologiczna, Legnica
  - Szpital Im. Kardynała Stefana Wyszyńskiego, Oddział Urologii, Lublin
  - Katedra i Klinika Urologii Pomorskiej Akademii Medycznej, Szczecin
  - Wojewódzki Szpital Specjalistyczny im. Janusza Korczaka, Oddział Urologii, Słupsk
  - Szpital Specjalistyczny, Oddział Urologii, Wejherowo
  - Katedra i Klinika Urologii AM we Wrocławiu, Wroclaw
  - Katedra i Klinika Urologii Śląskiej Akademii Medycznej, Zabrze
  - NZOZ Lekarze Urolodzy, Marek Rozniecki i Partnerzy, Łask